CLINICAL TRIAL: NCT06291623
Title: Molecular Analysis of Intracanal Microbes After Chemomechanical Procedure and Root Canal Medication: A Randomized Controlled Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Molecular Analysis
Record Dates: First submitted 2024-02-14; First posted 2024-03-04 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2024-01

CONDITIONS: Bacterial Viability of Necrotic Pulp With Asymptomatic Apical Periodontitis
Keywords: Dna , Rna extraction
MeSH Terms: interventions — Glycyrrhizic Acid; Calcium Hydroxide

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pre disinfection (30% H2O2, followed by 2.5% NaOCl) NaOCl inactivated with 5% sodium thiosulfate. (Experimental): sample was taken before pre disinfection protocol (30% H2O2, followed by 2.5% NaOCl) NaOCl will be inactivated with 5% sodium thiosulfate.
  Interventions: Drug: Glycyrrhizin
- Post disinfection (30% H2O2, followed by 2.5% NaOCl) NaOCl inactivated with 5% sodium thiosulfate. (Experimental): sample was taken after pre disinfection protocol, to check the sterility of the disinfected tooth surface and access
  Interventions: Drug: Glycyrrhizin
- Group 1 (n = 10): Ca(OH)2 (Experimental): 3 samples was taken before and after the treatment. Sample 1 was taken before Chemomechanical procedures Sample 2 was taken immediately after Chemomechanical procedures, intracanal medication was placed for 1 week Sample 3 was taken immediately after intracanal medication was removed
  Interventions: Drug: Glycyrrhizin
- Group 2 (n = 10): Glycyrrhizin (Experimental): 3 samples was taken before and after the treatment. Sample 1 was taken before Chemomechanical procedures Sample 2 was taken immediately after Chemomechanical procedures, intracanal medication was placed for 1 week Sample 3 was taken immediately after intracanal medication was removed
  Interventions: Drug: Glycyrrhizin

INTERVENTIONS:
Drug: Glycyrrhizin — used as intracanal medication for one week
  Other Names: Calcium hydroxide

SUMMARY:
This study aimed to evaluate clinically the intracanal microbes at molecular level after using established root canal medicament Calcium hydroxide and potential root canal medicament Glycyrrhizin.and Decontamination Analysis of Controls samples.

DETAILED DESCRIPTION:
Bacteria and their by-products are the main etiologic factors for pulpal and periapical diseases. The goals of endodontic treatment are to achieve complete disinfection and prevent reinfection in the root canal system and periapical tissues. Sterilization of root canals is limited by the presently available techniques, instruments, irrigants and intracanal medication. Thus, the focus should be on reducing intracanal bacterial populations to levels that are compatible with periapical tissue healing.Because root canal medicaments can come in contact with periapical tissue, in addition to having good antibacterial ability, they must also be biocompatible. In selecting root canal medicaments, it is necessary to consider their therapeutic benefits against their potential cytotoxic effects. Ideal root canal medicaments should have strong antibacterial properties and minimal cytotoxic effect on the host tissues.Globally, plants and their products are used for improving health. Plant extracts contain bioactive compounds like polyphenols, flavonoids, and many other compounds and chemical substances which play important roles to treat diseases. Due to health benefits, phytochemicals from plants generate a lot of interest, demanding further scientific evaluation.Glycyrrhiza which is known as licorice belonging to the Fabaceae, is native to southern Europe and parts of Asia . Glycyrrhizin has been labelled Generally Recognized as Safe (GRAS) by United States Food and Drug Administration (FDA) and has been considered safe for human consumption.Licorice roots have been used as a remedy for cough, laxative, menopausal hot flashes, peptic ulcer, and viral diseases . Licorice contains more than 20 triterpenoids and nearly 300 flavonoids. Among them, glycyrrhizin, 18 β-glycyrrhetinic acid, liquiritigenin, licochalcone A, licochalcone E and glabridin are the main active components which possess antimicrobial, antioxidant and anti-inflammatory activities.Evaluation of intra canal Bacterial levels and species before and after Chemomechanical procedures have been extensively explored by both culture (phenotype) and molecular techniques (genotype) . The latter became choice methods to assess persistent endodontic bacteria because of their high sensitivity and the ability to detect as-yet-uncultivated/difficult-to-culture bacteria.

ELIGIBILITY:
Inclusion Criteria:

Single-rooted teeth with a single canal, necrotic pulp (did not respond to sensitivity testing) and symptomatic apical periodontitis

* The age ranges from 19 to 60 years

Exclusion Criteria:- Receiving antibiotic treatment within the preceding 3 months.

* Reporting systemic disease.
* Teeth that could not be isolated with rubber dam.
* Teeth with periodontal pockets deeper than 3 mm.
* Root fracture or badly decayed teeth.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
minimizing of viable bacteria which showed by Real time PCR | after one week
  viable bacteria minimizing of Necrotic single canal with asymptomatic apical periodontitis

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahliya, Egypt